CLINICAL TRIAL: NCT00830921
Title: A Randomised Crossover Study to Investigate the Effect of Transcranial Magnetic Stimulation of the Anterior Cingulate Cortex on "Air Hunger"
Brief Title: Does Transcranial Magnetic Stimulation of the Cingulate Cortex Modulate the Perception of Dyspnoea?
Acronym: TMS
Status: Terminated | Type: Observational
Why Stopped: Lack of patients
Sponsor: University of Oxford (Other)
Responsible Party: Sponsor
Other Study IDs: 07/Q1607/48
Record Dates: First submitted 2009-01-27; First posted 2009-01-28 (Estimated); Last update posted 2012-06-18 (Estimated); Status verified 2012-06

CONDITIONS: Malignancy
Keywords: Histocytologically proven thoracic malignancy
MeSH Terms: conditions — Neoplasms | interventions — Transcranial Magnetic Stimulation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- 1: Patients will be identified from the Oxford Pleural Clinic and from referrals within the multi-disciplinary team including palliative care and oncology services.
  Screening criteria are based on normal practice and consecutive eligible patients will be offered trial entry. The principal investigator or a nominated member of staff will approach participants who fulfil the criteria for inclusion in the study. Screening logs will be kept.
  Interventions: Device: Transcranial Magnetic Stimulation

INTERVENTIONS:
Device: Transcranial Magnetic Stimulation — Transcranial magnetic stimulation (TMS) is a non-invasive method for altering brain activity in vivo.

SUMMARY:
The treatment we are studying is Transcranial Magnetic Stimulation (TMS). In TMS, an electromagnetic pulse is passed into the brain through a coil placed on the head. Previous studies have shown TMS to be capable of altering brain activity in specific areas; for example it has been used to improve mood in clinical depression. In this study we will assess if, by targeting TMS to the brain area responsible for feeling breathless, participants' breathlessness will be improved

DETAILED DESCRIPTION:
This protocol describes an exploratory crossover pilot study to assess whether targeted repetitive pulse Transcranial Magnetic Stimulation (TMS) i.e. targeted at the anterior cingulate cortex (ACC), affords relief of 'air hunger' in patients with breathlessness refractory to maximal medical therapy, compared to 'control' TMS directed at a remote site independent of the area of interest (within the lateral right parietal region of the brain).

12 right-handed patients suffering from refractory dyspnoea will receive pulses of targeted TMS or control TMS (crossover design), in a random order. The order will be random and use a minimisation procedure for baseline dyspnoea severity and sex. Repetitive targeted TMS (or control) pulses at 110% motor threshold at a frequency of 1Hz will be given for a 15 minute period1.

On a second, later, day the same subjects will perform the same protocol after receiving inhaled menthol or control (normal, non odorous air), in random order.

Outcomes will be assessed during the 10 minutes after targeted TMS/control TMS during which post stimulation inhibition of neural activity is expected.

ELIGIBILITY:
Inclusion Criteria:

1. Refractory dyspnoea (persisting sensation of air hunger despite optimisation of medical treatment)
2. Histocytologically proven thoracic malignancy
3. Written informed consent

Exclusion Criteria:

1. Age <18 years
2. Left-handed
3. Structural brain disease (including cerebral metastasis)
4. Personal or family history of seizures
5. Implantable metallic objects e.g. a pacemaker, or other contraindication to transcranial magnetic stimulation
6. Pregnant or breast feeding
7. Previous electroconvulsive therapy (ECT)
8. Poor mobility
9. Visual impairment
10. Lack of social support / home to go to after the study treatment
11. Alcohol dependency
12. PaCO2 >6kPa at rest
13. Inability to provide informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients attending out-patient clinic
Sampling Method: Probability Sample
Enrollment: 12 (Estimated)
Dates: Start 2008-02; Study Completion 2012-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Robert Davies, Study Director — Oxford Centre For Respiratory Medicine
Locations (1):
- Oxford Centre for Respiratory Medicine, Oxford, United Kingdom